CLINICAL TRIAL: NCT04283825
Title: The Therapeutic Efficacy of Psychological and Physical Rehabilitation Based Humanistic Care in Patients With Coronavirus Disease 2019
Brief Title: Humanistic Care in Patients With Coronavirus Disease 2019
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: We cannot enroll enough participants.
Sponsor: Second Affiliated Hospital of Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: XJTU2H-WH1
Record Dates: First submitted 2020-02-22; First posted 2020-02-25 (Actual); Last update posted 2020-03-17 (Actual); Status verified 2020-02

CONDITIONS: Coronavirus Disease 2019
Keywords: coronavirus disease 2019; physical rehabilitation; psychological rehabilitation
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Humanistic care (Experimental): In addition to routine therapy, the combinations of different psychological and physical rehabilitation activities will be applied to the patients.
  Interventions: Behavioral: Psychological and physical rehabilitation based humanistic care
- Non-humanistic care (No Intervention): Patients only receive routine therapy.

INTERVENTIONS:
Behavioral: Psychological and physical rehabilitation based humanistic care — This Psychological and physical rehabilitation based humanistic care regimen is generated from the experience of the National medical team members in Wuhan, from our hospital. In addition to the routine therapy, we will apply this comprehensive humanistic care regimen to the patients according to their condition. The patients will be stratified by the severity and receive different combinations of Psychological and physical rehabilitation activities.
  Arms: Humanistic care

SUMMARY:
As of February 17th, 2020, China has 76396 confirmed cases of coronavirus disease 2019 (COVID-19), including 2348 deaths. Although the impact factors of clinical outcomes among hospitalized patients still need to be clarified, some of the therapeutic regimens have shown the potency in the treatment of severe cases. Investigators aim to evaluate the efficacy of psychological and physical rehabilitation based humanistic care in the treatment of COVID-2019.

DETAILED DESCRIPTION:
As of February 17th, 2020, China has 76396 confirmed cases of coronavirus disease 2019 (COVID-19), including 2348 deaths. Although the impact factors of clinical outcomes among hospitalized patients still need to be clarified, some of the therapeutic regimens have shown their potency in the treatment of severe cases. Investigators aim to evaluate the efficacy of psychological and physical rehabilitation based humanistic care in the treatment of COVID-2019. As the national medical team sent to Wuhan, investigators proposed a Psychological and physical rehabilitation based humanistic care regimen generated from our experience in treating patients with COVID-2019. In addition to routine therapy, investigators will apply this comprehensive humanistic care regimen to the patients according to their condition to see the efficacy to this regimen.

ELIGIBILITY:
Inclusion Criteria:

* Inpatients with 2019 Novel Coronavirus infection

Exclusion Criteria:

* Patients can not follow-up;
* Investigator considering inappropriate.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-02-22 (Estimated); Primary Completion 2020-04-30 (Estimated); Study Completion 2020-05-15 (Estimated)

PRIMARY OUTCOMES:
Recovery Time | 1 month
  Time for recovery from admission to discharged

SECONDARY OUTCOMES:
Self-rating depression scale | 1 month
  Self-rating depression scale will be finished from patients by a scale table designed by investigator
Survival rate | 1 month
  Survival rate of the patient after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Shouping Gong, MD, PhD, Principal Investigator — Second Affiliated Hospital of Xi'an Jiaotong University

IPD SHARING:
Plan to Share IPD: No